CLINICAL TRIAL: NCT04987866
Title: Vibration Anesthesia for Propofol- Rocuronium Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E1-21-1740
Record Dates: First submitted 2021-07-01; First posted 2021-08-03 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-04

CONDITIONS: Vibration; Pain Due to Certain Specified Procedures
Keywords: vibration; analgesia; propofol injection pain; rocuronium injection pain
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group Vibration (Experimental): The participants who were chose an opaque envelope containing yellow paper represented the vibration group (Group V). After 1 min of pre-treatment with the vibration device on the intravenous catheter trace, we manually injected 2-2,5 mg/kg, 1% propofol (Propofol 1%, Fresenius 20 ml flacon, Germany) over 15 s. Observer rated the pain responses according to a four-point scale which developed by McCrirrick and Hunterand. Also asked the patients whether they had any discomfort. After the propofol injection, pain scores were observed during propofol injection and 20 seconds after the injection, and hemodynamic records were taken. 0,6 mg/kg rocuronium (Esmeron® 50 mg.5ml-1 N.V. Organon, Oss, Holland) were injected over 10 seconds. The movement response to rocuronium injection pain was evaluated by the same observer on a four-point scale (FPS) during and after 20 seconds rocuronium injection.
  Interventions: Device: vibration device , Beauty bar facial massaging device, T-Shape Electric Sign Face Massage Tools, Dangshan, China
- group Control (No Intervention): The participants who were chose an opaque envelope containing red paper represented the group control (Group C).Only propofol and rocuronium were given to these patients. propofol injection made manually 2-2,5 mg/kg, 1% propofol (Propofol 1%, Fresenius 20 ml flacon, Germany) over 15 s. Patients were observed during and after the injection of propofol for 20 seconds. Observer rated the pain responses according to a four-point scale which developed by McCrirrick and Hunter. During the injection of propofol, we also asked the patients whether they had any discomfort. After the propofol injection for 20 seconds, pain scores were observed, and hemodynamic records were taken. 0,6 mg/kg rocuronium (Esmeron® 50 mg.5ml-1 N.V. Organon, Oss, Holland) were injected over 10 seconds. The movement response to rocuronium injection pain was evaluated by the same observer on a four-point scale (FPS) during and 20 seconds after the rocuronium injection.

INTERVENTIONS:
Device: vibration device , Beauty bar facial massaging device, T-Shape Electric Sign Face Massage Tools, Dangshan, China — The vibration device is a reusable, handheld device with a battery-powered motor and a vibration frequency of approximately 6000 times per minute (Beauty bar facial massaging device, T-Shape Electric Sign Face Massage Tools, Dangshan, China)
  Arms: group Vibration

SUMMARY:
Despite numerous strategies for preventing or alleviating pain associated with propofol and rocuronium injections, it remains common and distressing for patients. Vibration is an effective method of reducing pain during facial cosmetic injections and some venipuncture procedures. But it has not been previously studied in the context of propofol or rocuronium injection pain. This randomized study aims to evaluate the effect of vibration anesthesia on the incidence and severity of propofol and rocuronium injection pain.

DETAILED DESCRIPTION:
Due to their rapid onset and short duration of action, ease of titration, recovery, and favorable profile for side effects, propofol and rocuronium are agents frequently used together in anesthesia practice and for rapid-sequence intubation. However, both cause severe discomfort due to pain in the injection arm. Some patients recall the induction of anesthesia as the most painful part of the perioperative period.

Vibration anesthesia has repeatedly been shown to alleviate pain sensation effectively and safely. Vibration anesthesia device is designed to reduce the pain from minor procedures, such as injection of medications, suture or staple removal, phlebotomy and even venipuncture pain in pediatric patients. The advantages of this device include its low cost, lack of adverse effects, and ease of use.

It has been shown to reduce pain with a mechanism based on the gate control theory, which states that vibrations stimulate the dorsal horn neurons, the sites at which pain signals are modulated and thus block full transmission of the pain.The investigators therefore proposed this randomized controlled study to compare the effectiveness of a vibration device for propofol and rocuronium injection pain during general anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Patients who are planned to undergo gynecology operations

Exclusion Criteria:

* Participants who were pregnant,
* Patients who had a recent history of a severe allergic or hypersensitivity reaction to propofol or rocuronium

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
preventing or reducing propofol injection pain | patients were observed during and after the injection of propofol for 20 seconds by an observer
  Observer rated the pain responses according to a four-point scale. After the injection of propofol to, we also asked the patients whether they had any discomfort.The severity of propofol- injection was evaluated using the following four-point pain response scale developed by McCrirrick and Hunter: level 0: (no pain) no verbal/ facial/ motor reaction to the injection; level 1: (mild pain) a minor verbal/ facial/ motor reaction to the injection but no physical activity or wrist joint movements; and level 2: (moderate pain), pain when asked by the anesthesiologist, or complaint of pain during the injection accompanied by physical activity- facial grimacing or withdrawal of the arm (elbow-shoulder); and level 3: (sever pain), a response accompanied by a facial expression of pain, or a strong vocal response, tears, arm withdrawal, and full body reaction ( including other body movements)
preventing or reducing rocuronium injection pain | patients were observed during and after the injection of rocuronium for 20 seconds by an observer
  The movement response to rocuronium injection pain was evaluated by the same observer on a four-point scale (FPS). The scale was 0: no movement, 1: movement only the wrist, 2: movement of only the arm (elbow-shoulder) and, 3: general response, movement more than one extremity. 2 minutes after induction, intubation was completed.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No